CLINICAL TRIAL: NCT01731496
Title: Improving Communication and Health for Adolescents With Technology - Implementation of Immunization Strategy
Brief Title: The Efficacy of Reminders to Complete HPV Series
Acronym: ICHAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Cynthia Rand, Associate Professor, Pediatrics, University of Rochester
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Health Services Research
Other Study IDs: 5K08HS017951-03 (AHRQ)
Record Dates: First submitted 2012-11-15; First posted 2012-11-21 (Estimated); Last update posted 2015-02-06 (Estimated); Status verified 2015-02

CONDITIONS: Completion of Three Dose Series of HPV; Improvement in Vaccine Intervals Between HPV Doses
Keywords: Human Papillomavirus

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Telephone reminder (Experimental): Telephone message reminder to parents of adolescents whose child is due for a 2nd or 3rd dose of HPV vaccine.
  Interventions: Other: Telephone reminder
- Text Message reminder (Experimental): Text message reminder to parents of adolescents whose child is due for a 2nd or 3rd dose of HPV vaccine.
  Interventions: Other: Text Message reminder
- Control: Telephone (No Intervention)
- Control: Text Message (No Intervention)

INTERVENTIONS:
Other: Telephone reminder — One week prior to when a child is due for either their 2nd or 3rd HPV vaccine, their parent will receive a telephone reminder to call to make an appointment to receive their next dose. A total of 3 reminders will be sent.
  Arms: Telephone reminder
Other: Text Message reminder — One week prior to when a child is due for either their 2nd or 3rd HPV vaccine, their parent will receive a text message reminder to call to make an appointment to receive their next dose. A total of 3 reminders will be sent.
  Arms: Text Message reminder

SUMMARY:
The human papillomavirus (HPV) vaccine is routinely recommended for both adolescent girls and boys starting at age 11, although it can be offered as young as 9 years of age. This is a 3-dose series and many adolescents do not complete it after getting the first dose. This study will study how effective it will be to send reminders to parents to schedule an appointment when their child is due for the next dose of HPV. Parents can chose whether they would like a phone call or text message reminder. This study will determine if the reminders work, and if one method is better than another (phone message vs. text message).

ELIGIBILITY:
Inclusion Criteria:

* Parents of adolescents aged 10 - 17 who have had at least 1 dose of HPV
* Patients aged 18 - 21 who have had at least 1 dose of HPV

Exclusion Criteria:

Ages: 10 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 749 (Actual)
Dates: Start 2012-04; Primary Completion 2014-05 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
HPV completion rate | One Year
  Post intervention HPV vaccination rates will be summarized by intervention group with frequencies and proportions, and will be compared between groups using chi square or Fisher's exact test as appropriate

SECONDARY OUTCOMES:
HPV Dosing Intervals | One Year
  Dosing intervals will be summarized by group with mean, median, standard deviation and will be compared between groups using a two sample t-test.

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Rand, MD, MPH, Principal Investigator — University of Rochester
Locations (3):
- United States (3):
  - Culver Medical Group, Rochester, New York
  - Highland Family Medicine, Rochester, New York
  - Strong Pediatric Practice, Rochester, New York

REFERENCES:
- [Derived] Rand CM, Vincelli P, Goldstein NPN, Blumkin A, Szilagyi PG. Effects of Phone and Text Message Reminders on Completion of the Human Papillomavirus Vaccine Series. J Adolesc Health. 2017 Jan;60(1):113-119. doi: 10.1016/j.jadohealth.2016.09.011. Epub 2016 Nov 8. PMID 27836533